CLINICAL TRIAL: NCT06454630
Title: A Phase 2, Multicenter, Randomized, Open-Label, Active Control Study of REGN7508, a Factor XI Monoclonal Antibody, for Prevention of Venous Thromboembolism After Elective, Unilateral, Total Knee Arthroplasty (ROXI-VTE II)
Brief Title: A Trial to Learn How Well REGN7508 Works for Preventing Blood Clots After a Knee Replacement in Adult Participants
Acronym: ROXI-VTE II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R7508-DVT-2360; 2023-508602-14-00 (Other: EU CT Number)
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Venous Thromboembolism
Keywords: Anti-factor XI (FXI) monoclonal antibody; Venous thromboembolism (VTE); Unilateral total knee arthroplasty (TKA)
MeSH Terms: conditions — Venous Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- REGN7508 (Experimental)
  Interventions: Drug: REGN7508
- Enoxaparin (Active Comparator)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: REGN7508 — Administered by single intravenous (IV) dose
  Arms: REGN7508
Drug: Enoxaparin — Administered by subcutaneous (SC) dose daily through the time of venography (or day 12, whichever is earlier)
  Other Names: Inhixa
  Arms: Enoxaparin

SUMMARY:
This study is researching an experimental drug called REGN7508 (called "study drug"). The study is focused on adults undergoing elective, unilateral (one side) total knee replacement (TKR) surgery.

The aim of the study is to see how effective the study drug is at preventing venous thromboembolism (VTE) and other related diseases after unilateral total knee replacement surgery.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Undergoing a primary elective unilateral TKA
2. Has a body weight ≤130 kg at screening visit
3. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and electrocardiograms (ECG's) performed at screening and/or prior to administration of initial dose of study drug as described in the protocol
4. Is in good health based on laboratory safety testing obtained during the screening period as described in the protocol

Key Exclusion Criteria:

1. History of bleeding in the past 6 months prior to dosing requiring hospitalization or transfusion; history of intracranial or intraocular bleeding, excessive operative or post-operative bleeding, and traumatic spinal or epidural anesthesia; history of bleeding diathesis
2. History of thromboembolic disease or thrombophilia
3. History of major surgery, including brain, spinal, or ocular, within approximately the past 6 months
4. History of major trauma within approximately the past 6 months prior to dosing
5. Hospitalized (>24 hours) for any reason within 30 days of the screening visit
6. Has an estimated glomerular filtration rate (GFR) of <45 mL/min/1.73m^2 at the screening visit using one of the following formulas: the Modification of Diet in Renal Disease (MDRD) equation, the Chronic Kidney Disease Epidemiology Collaboration equation, or equivalent equation

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Incidence of confirmed, adjudicated VTE | Through day 12

SECONDARY OUTCOMES:
Incidence of major bleeding | Up to approximately Day 12
Incidence of clinically relevant non-major (CRNM) bleeding | Up to approximately Day 12
Incidence of treatment emergent adverse events (TEAEs) | Through end of study; approximately Day 75
Incidence of major VTE | Through day 12
Incidence of Deep venous thrombosis (DVT) | Approximately Day 12
Concentrations of REGN7508 in serum | Through end of study; approximately Day 75
Change in activated partial thromboplastin time (aPTT) | Baseline to end of study; approximately Day 75
Change in prothrombin time (PT) | Baseline to end of study; approximately Day 75
Incidence of anti-drug antibodies (ADA) to REGN7508 | Through end of study; approximately Day 75
Titer of ADA to REGN7508 | Through end of study; approximately Day 75

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (14):
- Bulgaria (2):
  - Multi-profile Hospital for Active Treatment Hearth and Brain EAD, Pleven
  - Multiprofile Hospital For Active Treatment Park Hospital Ltd., Plovdiv
- Hungary (2):
  - Budai Irgalmasrendi Korhaz, Budapest
  - Szolnoki MAV Hospital, Szolnok
- Latvia (5):
  - Vidzemes Hospital, Valmiera, Valmieras Aprinkis
  - Liepaja Regional Hospital, Liepāja
  - Riga's 2nd Hospital, Riga
  - Hospital of Traumatology and Orthopaedics, Riga
  - Orto Klinika, Riga
- Lithuania (3):
  - Lietuvos sveikatos mokslu universiteto ligonine Kauno klinik, Kaunas, Kaunas County
  - Lithuanian University of Health Sciences Kaunas Hospital, Kaunas
  - Klaipeda University Hospital, Klaipėda
- Poland (2):
  - Specjalistyczny Szpital im. E. Szczeklika w Tarnowie, Tarnów, Lesser Poland Voivodeship
  - Clinic of Orthopaedics and Paediatric Orthopaedics, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry),
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Weitz JI, Kithcart AP, O'Brien MP, Levy O, Marin E, Onisko M, Mohammadi KA, Li D, Meagher KA, Chang HH, Olenchock BA, Gutstein DE, Segers A, Roberts RS, Bonaca MP, Raskob GE. Efficacy and safety of REGN9933A2 and REGN7508Cat for preventing postoperative venous thromboembolism (ROXI-VTE-I and ROXI-VTE-II): two randomised, open-label, phase 2 trials. Lancet. 2025 Nov 29;406(10519):2551-2563. doi: 10.1016/S0140-6736(25)02097-5. Epub 2025 Nov 8. PMID 41218619